CLINICAL TRIAL: NCT00675272
Title: Organ Donation and Vasopressor Use: Effects of Hydrocortisone Treatment
Brief Title: Organ Donation and Hydrocortisone Treatment
Acronym: HYDRO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Routine use of corticoids became standard therapy
Sponsor: Kuopio University Hospital (Other)
Collaborators: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Stepani Bendel, MD PhD, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KUH5070197
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Brain Death
Keywords: brain death; subarachnoid hemorrhage; traumatic brain injury; brain injury; intracerebral hemorrhage; organ donation
MeSH Terms: conditions — Brain Death; Subarachnoid Hemorrhage; Brain Injuries, Traumatic; Brain Injuries; Cerebral Hemorrhage | interventions — Hydrocortisone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): hydrocortisone treatment 50mg iv x4
  Interventions: Drug: hydrocortisone
- 2 (Placebo Comparator): Placebo iv every 6 hours
  Interventions: Drug: sodium chloride

INTERVENTIONS:
Drug: hydrocortisone — hydrocortisone 50mg iv. every 6 hours
  Arms: 1
Drug: sodium chloride — sodium chloride every 6 hours iv
  Arms: 2

SUMMARY:
Brain death patients who are selected for organ donation very often suffer from haemodynamic instability. To treat this, high amounts of vasoactive drugs(norepinephrine) may be needed to raise blood pressure. However,norepinephrine may have negative influence on several organs causing reduced blood flow ischemia. Our hypothesis is that hydrocortisone treatment may reduce the amount of vasoactive drugs needed to keep the blood pressure stable in patients selected for organ donation.

DETAILED DESCRIPTION:
When patients are treated in the ICU only as possible organ donators they will be assessed for eligibility for the study. Iv hydrocortisone or placebo will be administered every 6 hours. Several hormonal samples will be collected.

ELIGIBILITY:
Inclusion Criteria: all have to be fulfilled

* severe brain injury or subarachnoid hemorrhage which progrediates to brain death and patients are treated only as candidates for organ donation in the ICU
* no other reasons for treatment than organ donation
* informed consent from official representative

Exclusion Criteria:

* age under 18
* pregnancy
* corticoid treatment before study entry
* adrenal insufficiency
* hypophyseal insufficiency
* treatment with etomidate one week before study entry
* participating in an other study
* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-05; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
dosage and time on norepinephrine treatment | in ICU

SECONDARY OUTCOMES:
Hormone levels and number of organs donated | Hospital treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stepani Bendel, MD, Study Director — Kuopio University Hospital; Esko Ruokonen, MD, PhD, Study Director — Kuopio University Hospital; Jyrki Tenhunen, MD, PhD, Study Chair — Tampere UH; Anna-Maija Antman, MD, Principal Investigator — Tampere UH
Locations (2):
- Finland (2):
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere